CLINICAL TRIAL: NCT05049122
Title: A Single-arm, 52 Weeks, Phase 4 Study to Assess the Efficacy and Safety of Dupilumab in Patients With Chronic Rhinosinusitis With Nasal Polyposis (CRSwNP) Who Are Not Adequately Controlled With Existing Therapies
Brief Title: Dupilumab in Japanese Patients With Chronic Rhinosinusitis With Nasal Polyp (SINUS-M52)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Sanofi (Industry)
Collaborators: Regeneron Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LPS16872
Record Dates: First submitted 2021-09-14; First posted 2021-09-17 (Actual); Results first posted 2024-01-22 (Actual); Last update posted 2025-09-11 (Actual); Status verified 2025-09

CONDITIONS: Chronic Rhinosinusitis With Nasal Polyps
MeSH Terms: interventions — dupilumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Dupilumab (Experimental): Dupilumab every 2 weeks (q2w). Dosing interval may be changed from q2w to q4w at week 24
  Interventions: Drug: Dupilumab SAR231893

INTERVENTIONS:
Drug: Dupilumab SAR231893 — Pharmaceutical form: solution for injection Route of administration: subcutaneous (SC)
  Other Names: REGN668

SUMMARY:
This was a Phase 4, open-label, single-arm, multicenter study to evaluate the efficacy and safety of dupilumab subcutaneous (SC) injection monotherapy in Japanese participants aged 18 or older with CRSwNP that is not adequately controlled with existing therapies.

Duration of study period (per participant):

* Screening Period (2 to 4 weeks)
* Intervention Period (up to 52 weeks±3 days)

ELIGIBILITY:
Inclusion Criteria:

* Participants ≧18 years of age.
* Participants with bilateral sinonasal polyposis that despite prior treatment with systemic corticosteroids (SCS) anytime within the past 2 years; and/or had a medical contraindication / intolerance to SCS; and/or had prior surgery for NP at the screening visit, had:

  * An endoscopic bilateral NPS of at least 5 out of a maximum score of 8 (with a minimum score of 2 in each nasal cavity).
  * Ongoing symptoms (for at least 8 weeks prior to Visit [V] 1) of nasal congestion/blockage/obstruction with moderate or severe symptom severity (score 2 or 3) at V1 and a weekly average severity of greater than 1 at the time of enrollment (V2), and loss of smell, rhinorrhea (anterior/posterior).
* Participant's body weight > 30 kg at V1.
* Signed written informed consent.

Exclusion Criteria:

* Participant with conditions/concomitant diseases making them non evaluable at V1 or for the primary efficacy endpoint such as: Antrochoanal polyps; Nasal septal deviation that would occlude at least one nostril; Acute sinusitis, nasal infection or upper respiratory infection; Ongoing rhinitis medicamentosa; Eosinophilic granulomatosis with polyangiitis (Churg-Strauss syndrome), granulomatosis with polyangiitis (Wegener's granulomatosis), Young's syndrome, Kartagener's syndrome or other dyskinetic ciliary syndromes, concomitant cystic fibrosis; Radiologic suspicion, or confirmed invasive or expansive fungal rhinosinusitis;
* Participant with nasal cavity malignant tumor and benign tumors (eg, papilloma, blood boil, etc).
* Participant diagnosed with, suspected of, or at high risk of endoparasitic infection, and/or use of antiparasitic drug within 2 weeks before V1 or during screening
* Undergone any and/or sinus intranasal surgery within 6 months before V1.
* Participant who had participated in prior dupilumab clinical study or had been treated with commercially available dupilumab

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2021-10-22 (Actual); Primary Completion 2022-12-21 (Actual); Study Completion 2023-07-05 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Investigational site JAPAN, Japan, Japan

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org

REFERENCES:
- [Derived] Fujieda S, Takabayashi T, Ohta N, Yoshikawa M, Kibe Y, Ishida M, Suzuki K, Takahashi Y, Amin N, Wright L, Robinson L, Yahata K. Effectiveness and Safety of Dupilumab Monotherapy in Japanese Patients With Chronic Rhinosinusitis With Nasal Polyps. Laryngoscope. 2025 Dec;135(12):4625-4632. doi: 10.1002/lary.70037. Epub 2025 Aug 30. PMID 40884290
- See also: LPS16872 Plain Language Results Summary — https://www.trialsummaries.com/Study/StudyDetails?id=25292&tenant=MT_SNY_9011

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 9 centers in Japan. A total of 30 participants were screened from 22 Oct 2021 to 22 Jun 2022 of which 5 were screen failures due to not meeting eligibility criteria.
Pre-assignment Details: The study consisted of a screening period (up to 4 weeks) and a treatment period (up to 52 weeks). A total of 25 participants were enrolled in this study. The study duration for each participant was up to 56 weeks.
Groups:
- Dupilumab 300 Milligrams (mg): Participants received dupilumab 300 mg every 2 weeks (q2w) up to Week 24. Participants with stable disease (nasal polyp score [NPS] improvement from baseline to both Weeks 16 and 24 of greater than or equal to [>=]2 points) at Week 24 received dupilumab 300 mg every 4 weeks (q4w) after Week 24 up to Week 48 and those who could not achieve stable disease at Week 24 continued to receive dupilumab 300 mg q2w after Week 24 up to Week 50. All participants were followed up to Week 52.
Period: Overall Study
Arm/Group | Dupilumab 300 Milligrams (mg)
Started (Enrolled) | 25
Participants Who Completed the Week 24 Study Treatment Period as Per Protocol | 23
Participants Who Were Considered Stable Condition at Week 24 | 3
q4w Regimen Participants (Stable Condition)Who Completed Week 52 Study Treatment Period Per Protocol | 3
Participants Who Continued the q2w Regimen | 20
The q2w Regimen Participants Who Completed the Week 52 Treatment Period as Per Protocol | 19
Completed (Participants who completed the Week 52 treatment period as per protocol) | 22
Not Completed | 3
Not completed — Adverse event not related to Coronavirus Diesease-2019 | 1
Not completed — Participant moved | 1
Not completed — At the direction of the doctor | 1

BASELINE CHARACTERISTICS:
Population: The Enrolled analysis set consisted of all participants with a treatment kit number allocated and recorded in the interactive response technology (IRT) database, regardless of whether the treatment kit was used or not.
Groups:
- Dupilumab 300 mg: Participants received dupilumab 300 mg q2w up to Week 24. Participants with stable disease (NPS improvement from baseline to both Weeks 16 and 24 of >=2 points) at Week 24 received dupilumab 300 mg q4w after Week 24 up to Week 48 and those who could not achieve stable disease at Week 24 continued to receive dupilumab 300 mg q2w after Week 24 up to Week 50. All participants were followed up to Week 52.
Arm/Group | Dupilumab 300 mg
Number analyzed (Participants) | 25
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.4 (13.56)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10
  Male | 15
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 25
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 0
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With NPS Improvement From Baseline >=1 at Week 24
Description: The NPS was the sum of right and left nostril scores as assessed by central video recordings of nasal endoscopy (NE). For each nostril, NPS was graded based on polyp size: Grade 0:No polyps; Grade 1:Small polyps in the middle meatus not reaching below the inferior border of the middle turbinate; Grade 2:Polyps reaching below the lower border of the middle turbinate; Grade 3:Large polyps reaching the lower border of the inferior turbinate or polyps medial to the middle turbinate; Grade 4:Large polyps causing complete obstruction of the inferior nasal cavity. Score ranged from 0-8; higher scores indicated more severity. The baseline value was defined as the last available value before first study treatment administration.
Time Frame: Baseline (Day 1) and Week 24
Population: The Per protocol (PP) analysis set consisted of all participants in modified intent-to-treat (mITT) set (Enrolled population with chronic rhinosinusitis with nasal polyp [CRSwNP] allocated to study treatment administered at least 1 dose of study treatment) and who did not receive intranasal corticosteroids (INCS) up to Week 24
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Dupilumab 300 mg
Number analyzed (Participants) | 25
percentage of participants | 92.0 [72.5 to 98.6]

2. Secondary Outcome: Change From Baseline in Bilateral NPS at Week 24
Description: The NPS was the sum of right and left nostril scores as assessed by central video recordings of NE. For each nostril, NPS was graded based on polyp size: Grade 0:No polyps; Grade 1:Small polyps in the middle meatus not reaching below the inferior border of the middle turbinate; Grade 2:Polyps reaching below the lower border of the middle turbinate; Grade 3:Large polyps reaching the lower border of the inferior turbinate or polyps medial to the middle turbinate; Grade 4:Large polyps causing complete obstruction of the inferior nasal cavity. Score ranged from 0-8; higher scores indicated more severity. For participants who discontinued for other reasons, missing data are imputed using multiple imputation techniques assuming missing at random, and non-missing data collected after treatment discontinuation were used in the analysis. The baseline value was defined as the last available value before first study treatment administration.
Time Frame: Baseline (Day 1) and Week 24
Population: The PP analysis set consisted of all participants in mITT allocated to study treatment administered at least 1 dose of study treatment, and who did not receive INCS up to Week 24.
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Dupilumab 300 mg
Number analyzed (Participants) | 25
score on a scale | -2.4 (0.34)

3. Secondary Outcome: Change From Baseline in Nasal Congestion/Obstruction (NC) Symptom Severity Score Using the CRSwNP Nasal Symptom Diary at Week 24
Description: The NC was assessed by the participant using a diary on a daily basis from Visit 1 and throughout the study on a 0 to 3 categorical scale (where 0 = no symptoms, 1 = mild symptoms, 2 = moderate symptoms and 3 = severe symptoms). It was scored as a reflective score (evaluation of symptom severity over the past 24 hours) by the participants. The score ranged from 0-3; higher scores indicated more severity. The baseline value was defined as the last available value before first study treatment administration. For participants who discontinued for other reasons, missing data are imputed using multiple imputation techniques assuming missing at random, and non-missing data collected after treatment discontinuation were used in the analysis. The baseline value was defined as the last available value before first study treatment administration.
Time Frame: Baseline (Day 1) and Week 24
Population: as for outcome 2
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Dupilumab 300 mg
Number analyzed (Participants) | 25
score on a scale | -1.58 (0.213)

4. Secondary Outcome: Change From Baseline in Opacification of Sinuses Assessed by Computerized Tomography (CT) Scan Using the Lund Mackay (LMK) Score at Week 24
Description: The LMK system is based on localization with points given for degree of opacification: 0 = normal, 1 = partial opacification, 2 = total opacification. These points were applied to the maxillary, anterior ethmoid, posterior ethmoid, sphenoid, and frontal sinus on each side. The osteomeatal complex (OC) was graded as 0 = not occluded or 2 = occluded. The total score was the sum of scores from each side and ranged from 0 (normal) to 24 (more opacified); higher score indicated more severe disease. For participants who discontinued for other reasons, missing data are imputed using multiple imputation techniques assuming missing at random, and non-missing data collected after treatment discontinuation were used in the analysis. The baseline value was defined as the last available value before first study treatment administration.
Time Frame: Baseline (Day 1) and Week 24
Population: as for outcome 2
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Dupilumab 300 mg
Number analyzed (Participants) | 25
score on a scale | -5.6 (0.91)

5. Secondary Outcome: Change From Baseline in Total Symptom Score (TSS) at Week 24
Description: The TSS was the sum of participant-assessed nasal symptom scores for nasal congestion and/or obstruction, decreased/loss of sense of smell and rhinorrhea (average of the non-missing anterior/posterior nasal discharge). On a daily basis from Visit 1 and throughout the study, participants used a diary to respond to the morning individual rhinosinusitis symptom questions using a 0 to 3 categorical scale (where 0 = no symptoms, 1 = mild symptoms, 2 = moderate symptoms and 3 = severe symptoms). Total score ranged from 0 (no symptoms) to 9 (severe symptoms). Higher score indicated more severe symptoms. For participants who discontinued for other reasons, missing data are imputed using multiple imputation techniques assuming missing at random, and non-missing data collected after treatment discontinuation were used in the analysis. The baseline value was defined as the last available value before first study treatment administration.
Time Frame: Baseline (Day 1) and Week 24
Population: as for outcome 2
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Dupilumab 300 mg
Number analyzed (Participants) | 25
score on a scale | -4.20 (0.582)

6. Secondary Outcome: Change From Baseline in Loss of Smell Symptom Severity Score Using the Nasal Symptom Diary at Week 24
Description: The severity of loss of smell was reported by the participants using the nasal symptom diary with a 0 to 3 categorical scale (where 0 = no symptoms, 1 = mild symptoms, 2 = moderate symptoms and 3 = severe symptoms), higher score indicated more severe symptoms. For participants who discontinued for other reasons, missing data are imputed using multiple imputation techniques assuming missing at random, and non-missing data collected after treatment discontinuation were used in the analysis. The baseline value was defined as the last available value before first study treatment administration.
Time Frame: Baseline (Day 1) and Week 24
Population: as for outcome 2
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Dupilumab 300 mg
Number analyzed (Participants) | 25
score on a scale | -1.37 (0.258)

7. Secondary Outcome: Change From Baseline in Visual Analogue Scale (VAS) for Rhinosinusitis at Week 24
Description: The VAS for rhinosinusitis was used to evaluate the total disease severity. Rhinosinusitis was divided into mild, moderate and severe based on total severity VAS score (0 to 10 centimeters [cm] where mild: VAS 0 to 3; moderate: VAS >3 to 7 and severe: VAS >7 to 10). The participants were asked to indicate on a VAS the answer to the question: "How troublesome are your symptoms of your rhinosinusitis?" The range of the VAS was from 0 (not troublesome) to 10 (worst thinkable troublesome), where higher score indicated worse disease. For participants who discontinued for other reasons, missing data were imputed using multiple imputation techniques assuming missing at random, and non-missing data collected after treatment discontinuation were used in the analysis. The baseline value was defined as the last available value before first study treatment administration.
Time Frame: Baseline (Day 1) and Week 24
Population: as for outcome 2
Measure: Mean (Standard Error); unit: cm
Arm/Group | Dupilumab 300 mg
Number analyzed (Participants) | 25
cm | -5.41 (0.622)

8. Secondary Outcome: Number of Participants With Treatment-Emergent Adverse Events (TEAEs), Treatment-Emergent Serious Adverse Events (TESAEs) and TEAEs Leading to Treatment Discontinuation at the End of 24-Week Treatment Period
Description: An Adverse Event (AE) was defined as any untoward medical occurrence in a participant temporally associated with the use of study treatment, whether or not considered related to the study treatment. TEAEs were defined as AEs that developed or worsened in grade or became serious during TE period which was defined as the period from the time of first dose of study treatment until the last visit in the study. Serious adverse events (SAE) were defined as any untoward medical occurrence that at any dose: resulted in death, was life-threatening, required inpatient hospitalization or prolongation of existing hospitalization, resulted in persistent or significant disability/incapacity, was a congenital anomaly/birth defect, was a medically important event. Data reported is till the end of 24-week treatment period.
Time Frame: From Baseline (Day 1) up to Week 24
Population: The Safety analysis set consisted of all participants allocated to study treatment and administered at least 1 dose of study treatment before Week 24.
Measure: Count of Participants; unit: Participants
Arm/Group | Dupilumab 300 mg
Number analyzed (Participants) | 25
Participants
  Any TEAE | 11
  Any TESAE | 1
  Any TEAE leading to treatment discontinuation | 0

ADVERSE EVENTS:
Time Frame: From first treatment administration up to Week 52
Description: The Safety analysis set consisted of all participants allocated to study treatment administered at least 1 dose of study treatment during the intervention period.
Arm/Group | Dupilumab 300 mg
All-Cause Mortality (participants affected / at risk) | 0/25
Serious Adverse Events (participants affected / at risk) | 2/25
Other Adverse Events (participants affected / at risk) | 10/25
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dupilumab 300 mg (N=25)
Suicide Attempt (Psychiatric disorders) | 1 (1)
Vestibular neuronitis (Infections and infestations) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dupilumab 300 mg (N=25)
Covid-19 (Infections and infestations) | 5 (5)
Nasopharyngitis (Infections and infestations) | 2 (2)
Seasonal Allergy (Immune system disorders) | 2 (2)
Injection Site Erythema (General disorders) | 2 (6)
Pyrexia (General disorders) | 2 (3)
Accidental Overdose (Injury, poisoning and procedural complications) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor supports publication of clinical trial results but may request that investigators temporarily delay or alter publications in order to protect proprietary information. The Sponsor may also require that the results of multicenter studies be published only in their entirety and not as individual site data.

DOCUMENTS (2):
  • Study Protocol (2021-05-11): https://cdn.clinicaltrials.gov/large-docs/22/NCT05049122/Prot_000.pdf
  • Statistical Analysis Plan (2023-01-16): https://cdn.clinicaltrials.gov/large-docs/22/NCT05049122/SAP_001.pdf